CLINICAL TRIAL: NCT01605786
Title: Phase I and IIa Trial for Assessment of Safety, Immunogenicity (Phase Ia) and Efficacy (Phase IIa) Against Sporozoite Challenge of P. Falciparum Pre-Erythrocytic and Blood Stage (PfPEBS-LSP) Malaria Vaccine Candidate
Brief Title: Trial for Malaria Vaccine Candidate, PfPEBS (P. Falciparum Pre-Erythrocytic and Blood Stage)
Acronym: PEBS-POC1
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vac4All (Industry)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other); Radboud University Medical Center (Other); European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pf PEBS-Ia-IIa; 2012-002294-54 (EudraCT Number)
Record Dates: First submitted 2012-05-18; First posted 2012-05-25 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Malaria
Keywords: Malaria; Plasmodium falciparum; vaccine; ADCI; sporozoite challenge; pre-erythrocytic; erythrocytic
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PEBS Low dose (Experimental)
  Interventions: Biological: Lyophilised PEBS synthetic protein (PfPEBS)
- PEBS High dose (Experimental)
  Interventions: Biological: Lyophilised PEBS synthetic protein (PfPEBS)
- Control (Active Comparator)
  Interventions: Other: Rehydragel™ HPA

INTERVENTIONS:
Biological: Lyophilised PEBS synthetic protein (PfPEBS) — PfPEBS, is a synthetic polypeptide corresponding to amino acids 3112 to 3244 (131 aa) from the Pf 11.1 antigen in 3D7 parasite sequence. It is presented as lyophilised product in multi-dose vials (containing 105 μg for 3 doses of 30 μg ), looking like amorphous white powder. The vaccine is produced by SYNPROSIS in France.
  The 5μg dose vaccine will be formulated extemporaneously in aluminium hydroxide adjuvant and given as a 2-dose schedule with a 28 day interval.
  Arms: PEBS Low dose
Biological: Lyophilised PEBS synthetic protein (PfPEBS) — PfPEBS-LSP, is a synthetic polypeptide corresponding to amino acids 3112 to 3244 (131aa) from the Pf 11.1 antigen in 3D7 parasite sequence. It is presented as lyophilised product in multi-dose vials (containing 105 μg for 3 doses of 30 μg ), looking like amorphous white powder. The vaccine is produced by SYNPROSIS in France.
  The 30 μg dose vaccine will be formulated extemporaneously in aluminium hydroxide adjuvant and given as a 2-dose schedule with a 28 day interval.
  Arms: PEBS High dose
Other: Rehydragel™ HPA — Aluminium hydroxide adjuvant is being used as the adjuvant for the vaccine and will be used as the comparator in the control group. Vac4all is using Rehydragel™ (Manufacturer Reheis Inc.) which is a highly active protein adsorbent specially compounded for use as a fluid adjuvant. It has low oxide content and is carefully controlled for Al2O3 content and protein binding capacity. It has a lower viscosity than competing adjuvants, which makes it easier to process and handle.
  Subjects in the control group will be administered a 0.5 ml injection in a 2-dose schedule at 28 days interval. Each injection will contain approximately 600 µg of Al(OH)3 per injected dose corresponding to 200 µg equivalent of Al3+, similar to the amount being administered in the vaccine group.
  Arms: Control

SUMMARY:
This study intends to test the hypothesis that the malaria antigen PfPEBS, manufactured as a synthetic protein and adjuvanted with aluminium hydroxide will be well-tolerated and immunogenic (Phase 1), functionally active against the erythrocytic stages (Phase 1) and efficacious (Phase 2) against the pre-erythrocytic stages in protecting against an artificial malaria challenge using Pf sporozoites in a healthy adult population.

DETAILED DESCRIPTION:
The study will enroll 36 healthy adult subjects (18-45 years) and randomize them in a double-blind manner into 3 arms of 12 subjects each; 2 of the arms will receive either 5μg or 30μg, both adjuvanted with aluminium hydroxide, given as a 2-dose schedule with a 28 day interval. The third arm of 12 subjects will act as controls, and they will receive aluminium hydroxide only injections.

If the safety and immunogenicity results permit, the subjects will be challenged with live mosquito challenge delivering P falciparum sporozoites to assess pre-erythrocytic vaccine efficacy.

The PfPEBS molecule has been found to have in vivo and in vitro functional activity against the two stages that are clinically significant for malaria namely the pre-erythrocytic stages (sporozoite and liver stages) and the erythrocytic stages.

The formulation is a simple combination of a synthetic protein of 131 amino acids adjuvanted with aluminum hydroxide, the adjuvant with the widest safety records.

The combined Phase 1/2a study is designed in order to achieve 3 co-primary objectives

1. Phase 1: To demonstrate safety and tolerability
2. Phase 1: To measure the activity against the asexual blood stage of the parasite which is only indirectly estimated by the functional activity of elicited antibodies in ADCI under in-vitro conditions
3. Phase 2: To demonstrate efficacy against liver stages by measuring the proportion of subject that are protected following a live sporozoite challenge.

The mechanisms of defenses differ for "liver stages" and "erythrocytic stages". Defenses against "liver stages" are strongly related to the secretion of interferon γ by CD4+Th1 cells, whereas for blood stages the defences depend on antibodies.

Preliminary studies have demonstrated that low antigen doses such as 5 or 2μg produce strong CD4+Th1- interferon γ secreting cells with low antibody titers, whereas higher antigen doses such as 30 or 50μg induce lower CD4 Th1 cell response and markedly higher antibody responses.

Therefore the choice of the two dose ranges for the Pf-PEBS clinical trial protocol is aimed at testing the two main efficacy objectives, one against "liver stages" with a low dose, the other against "the blood stages" with the higher dose.

The Sponsor for the two Phases is Vac4all. The funder for the Phase Ia is the EMVDA programme of the European Commission. The funder for the Phase IIa is Vac4all

ELIGIBILITY:
Inclusion Criteria:

* Male and female age > 18 and < 45 years
* Good general health based on history, physical en laboratory examination
* Available for and willingness to undergo a P. falciparum sporozoite infected mosquito challenge following the immunization course
* Resident in or near Lausanne for the duration of the study having 24h access to a mobile telephone
* Willingness to stay in special accommodation (hotel or equivalent) from day 5 up to one day after parasite positivity , or up to day 15 post EHMI
* Agreement to refrain from blood donation during the course of the study and afterwards
* Negative pregnancy test and the use of effective contraception during the whole study period if deemed appropriate
* Willingness to undergo an HIV test and other serologies
* Willingness to allow investigators to notify their general practitioner, if any, of participation in this trial
* Willingness to allow investigators to request medical information, relevant for participation in this trial, from their general practitioner, if any
* Written informed consent following proper understanding of the meaning and procedures of the Phase I and IIa parts of the trial
* Agreement to inform study doctor and to release medical information concerning contra-indications for participation in the study
* Willingness to undergo screening for drugs such as amphetamines, opiates and cocaine

Exclusion Criteria:

* Any history of malaria
* Known exposure to malaria in the previous 6 months, defined as a visit to a malaria endemic region. For practical purposes, all regions for which malaria chemoprophylaxis is advised by travel clinic are considered malaria endemic
* Planned to travel to endemic malaria areas during the study period
* Prior administration of an investigational malaria vaccine
* Administration of a vaccine or gammaglobulin not foreseen by the clinical trial protocol within 30 days prior to the first immunization and up to six months after the last immunization.
* Participation in any other clinical trial within 90 days prior to the onset of the trial or more than four clinical trials in the past year
* The use of chronic medication (defined as more than 14 days), especially immunosuppressive agents or antibiotics during the study period
* The use of chronic immunosuppressive drugs or other immune modifying drugs within three months of vaccination (inhaled and topical corticosteroids are allowed)
* Positive serological tests for P. falciparum (PEBS) ELISA and/or a positive P. falciparum whole parasite ELISA
* Known hypersensitivity to vaccine components
* History of severe reactions or allergy to mosquito bites
* Contra indications to Malarone® including treatment taken by the volunteers that interfere with Malarone® (e.g. concurrent use of medicines that prolong QT interval)
* History of allergic disease to or reactions likely to be exacerbated by any component of the vaccine
* Any confirmed or suspected immunosuppressive or immunodeficiency condition, including asplenia.
* History of diabetes mellitus or cancer (except basal cell carcinoma of the skin)
* History of >2 hospitalisations for invasive bacterial infections
* Symptoms, physical signs and laboratory values suggestive of systemic disorders, including renal, hepatic, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric and other conditions, which could interfere with the interpretation of the study results or compromise the health of the volunteers
* An estimated, ten year risk of fatal cardiovascular disease of ≥5%, as estimated by the Systematic Coronary Risk Evaluation (SCORE) system.
* History of arrhythmia or prolonged QT interval or other cardiac disease
* Positive history for cardiac disease in the 1st and 2nd degree relative < 50 years old
* Clinically significant abnormalities in electrocardiogram (ECG) at screening
* Body Mass Index < 18 kg/m2 or > 32 kg/m2
* Blood pressure > 150/90 in two measurements
* Seropositive for HIV, HBV or HCV
* Any clinically significant deviation from the normal range in biochemistry or haematology blood tests or in urine analysis.
* Volunteers unable to be closely followed for social, geographic or psychological reasons
* Previous history of drug or addiction to alcohol abuse interfering with normal social function during a period of one year prior to enrolment in the study
* Having not reached 10 correct responses to the knowledge questionnaire

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-05 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Adverse events following vaccination | Up to one year following first vaccination
  The safety and reactogenicity of the vaccine will be assessed by comparing the proportion and severity of expected and unexpected adverse events as well as serious adverse events (SAE) between groups.
Change from baseline of antibodies active in the ADCI assay | Within one year following first vaccination
  The vaccine antigen should induce adequate antibodies that are active in the ADCI assay, which measures parasite killing of erythrocytic stages of the malaria parasite by antibodies in Monocyte-dependant manner and is hypothesized to be able to provide protection against clinical malaria disease.
Parasitemia following mosquito challenge | From Day 4 up to Day 21 post challenge
  Subjects will be monitored for emergence of malaria parasites in the blood, using the gold standard of thick film slide microscopy, and rapid diagnostic testing, RT-PCR and LAMP. Treatment will be initiated as soon as subjects are parasitemic, defined as >1 parasites per 400 fields in a thick blood film, OR a positive RDT OR two positive RT-PCR OR one positive result with RT-PCR AND one positive result with LAMP OR two positive results with two different methods.

SECONDARY OUTCOMES:
Antibodies against synthetic PEBS | Within one year following first vaccination
  This will be measured by ELISA
Antibodies against parasite antigen | Within one year following first vaccination
  This will be measured by the following methods: whole parasite extract, ELISA, Western Blot, IFAT
PEBS Interferon-Gamma | Within one year following first vaccination
  This will be measured by ELISPOT

CONTACTS AND LOCATIONS:
Overall Officials: Pierre L Druilhe, MD, Study Director — Vac4All; Francois Spertini, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois (CHUV)
Locations (1):
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland